CLINICAL TRIAL: NCT05747898
Title: Cannula-based Versus Common Needle-based Subcision in the Treatment of Posttraumatic Atrophic Facial Scars: A Clinical Trial
Brief Title: Cannula-based Versus Needle-based Subcision for Posttraumatic Atrophic Facial Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed, Lecturer of Dermatology, Venereology, and Andrology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: subatrophic001
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Scar; Atrophy
MeSH Terms: conditions — Cicatrix; Atrophy

STUDY DESIGN:
Intervention Model Description: Each scar was split into two equal halves; the upper right half were treated using a cannula- based subcision approach, while the lower left half was treated using a common needle-based procedure
Who Masked: Outcomes Assessor
Masking Description: The assessor was blinded to the treatment applied to each half of the scar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannula arm (Active Comparator): the cannula's 18 gauge tip was pointed upward and approximately parallel to the skin's surface when it was put into the superficial dermis, 1-2 millimeters away from the targeted scar. In order to completely remove fibrous tissue from the superficial dermis, a lancing motion (linear inserting-withdrawing needle action) was utilized first.
  Interventions: Procedure: cannula- based subcision
- Needle arm (Active Comparator): The needle's 27 gauge tip was pointed upward and approximately parallel to the skin's surface when it was put into the superficial dermis, 1-2 millimeters away from the targeted scar. In order to completely remove fibrous tissue from the superficial dermis, a lancing motion (linear inserting-withdrawing needle action) was utilized first.
  Interventions: Procedure: common- needle based subcision

INTERVENTIONS:
Procedure: cannula- based subcision — Insertion of a needle into the base of a cutaneous scar to cut fibrous tissue and help new collagen formation.
  Arms: Cannula arm
Procedure: common- needle based subcision — Insertion of a cannula into the base of a cutaneous scar to cut fibrous tissue and help new collagen formation.
  Arms: Needle arm

SUMMARY:
This study aims to evaluate the effectiveness of cannula- based subcision versus common needle subcision in treatment of posttraumatic atrophic facial scars

DETAILED DESCRIPTION:
In addition to cosmetic issues, atrophic scars can lead to psychological issues like social isolation, low self-esteem, and embarrassment. Subcision (Subcutaneous incision-less surgery) has been used for years to treat a variety of skin depressions, including atrophic acne scars and other depressed scars. Numerous modifications have been made throughout time to this surgical method to make it easier and more efficient. Although needle subcision is a straightforward, simple, useful, and practical procedure, it has many side effects and the overall success in this procedure is mild to moderate. So, in this study we evaluated the effectiveness of cannula- based subcision versus common needle subcision in treatment of posttraumatic atrophic facial scars.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (> 20-years old) with posttraumatic facial scar

Exclusion Criteria:

* other types of scars (e.g; postacne scars), pregnancy, lactation, bleeding or coagulation disorders, liability for keloid formation, history of kobnerization, and patients with systemic diseases (cardiac, chronic renal diseases, chronic liver diseases, asthma and hypertension) at the time of recruitment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Vancouver scar scale (VSS) | 4 months
  The (VSS) examines vascularity, pliability, pigmentation, and height, yielding a total score that ranges from 0 to 14. The original rating system was as follows: Vascularity (0=normal, 1=pink, 2=red, 3=purple), Pliability (Normal=0, Flat=0, Supple=1, Yielding=2, Firm=3, Ropes=4, Contracture=5), Pigmentation (0=normal, 1=hypo-pigmentation, 2=mixed pigmentation, 3=hyper-pigmentation), and Height (Flat=0 <2 mm=1 2-5 mm=2 >5 mm=2) .

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Mohamed, MD, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt